CLINICAL TRIAL: NCT02720185
Title: Window of Opportunity Study of Dasatinib in Operable Triple Negative Breast Cancers With Nuclear Epidermal Growth Factor Receptor (nEGFR)
Brief Title: Window of Opportunity Trial of Dasatinib in Operable Triple Negative Breast Cancers With nEGFR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to COVID-19 related slow enrollment and funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UW15114; 1R01CA193004-01A1 (NIH); NCI-2016-00237 (Registry Identifier: NCI Trial ID); 2015-1578 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 8/29/2019 (Other: UW Madison)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2022-02-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Breast Neoplasms; Triple Negative Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib 100mg (Experimental): Dasatinib 100mg for 7-10 days until day prior to surgery
  Interventions: Drug: Dasatinib; Procedure: Conventional Surgery; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Dasatinib — 100mg oral once daily dasatinib taken for 7-10 days up to the day prior to planned surgery or research biopsy (neoadjuvant chemotherapy group)
  Other Names: 732517; 863127-77-9; BMS-354825; Sprycel
Procedure: Conventional Surgery — Undergo surgery
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Primary Objective:

To determine if dasatinib, an inhibitor of the Src family kinases, can prevent the nuclear translocation of the epidermal growth factor receptor (EGFR) in Stage I-III, nuclear EGFR positive, triple negative breast cancers (TNBC).

Secondary Objectives:

1. To examine the safety and tolerability of dasatinib in patients with operable TNBC
2. To explore potential intracellular mechanisms which impact dasatinib effect on cellular localization of EGFR in operable TNBC.
3. To examine the pathologic complete response (pCR) rates to standard neoadjuvant chemotherapy in nEGFR+ TNBC
4. To examine breast cancer recurrence rates and patterns of metastatic recurrent in nEGFR+ TNBC

ELIGIBILITY:
Inclusion Criteria for nEGFR testing:

* Patients must have histologically or cytologically confirmed Stage I-III triple negative breast cancer

  * estrogen receptor (ER) and progesterone receptor (PR) must be <1% by standard assay methods
  * human epidermal growth factor receptor-2 (HER2) must be either 0, 1+ by immunohistochemistry (if 2+, in situ hybridization method used to define HER2) OR have HER2: 17 centromere signal of <2.0 using a standard in situ hybridization method
* No prior therapy for current breast cancer
* Meet criteria for neoadjuvant chemotherapy or primary breast surgery, as determined by primary oncologist and surgeon

Inclusion Criteria for study therapy:

* nEGFR positive
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Patients must have normal organ and marrow function as defined below:
* leukocytes ≥3,000/mcL
* absolute neutrophil count ≥1,500/mcL
* platelets ≥150,000/mcL
* total bilirubin <1.25x institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
* creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 30 days after the final dose. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients not able to swallow oral medications or with gastrointestinal conditions that may impact absorption of dasatinib.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib.
* Patients receiving any medications or substances that are moderate or strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, medications should be reviewed by the UW Pharmacy Research Center for any contraindicated medications. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* H2 antagonists and proton pump inhibitors are not allowed
* Anticoagulants (ie. Coumadin, heparin, anti-Xa inhibitors) and anti-platelet agents (ie. aspirin) are not allowed. NSAIDS and acetaminophen are allowed on study.
* Medications known to prolong QTC are not allowed (See Appendix B)
* No history of prolonged QTC or cardiomyopathy unless normal QTC and ejection fraction confirmed within 1 month prior to study entry.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because dasatinib is a pregnancy category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated with dasatinib and not resumed until at least 2 weeks after the final dose.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dasatinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Contraindication to repeat breast biopsy (neoadjuvant chemotherapy group)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari B Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Illinois Hospital and Health Systems (Outpatient Care Center), Chicago, Illinois
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were entered on study at the University of Wisconsin Carbone Cancer Center. Participants were enrolled from May 2017 to June 2020.
Period: Overall Study
Arm/Group | Dasatinib 100mg
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib 100mg
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2
  40-49 years | 1
  50-59 years | 1
  60-69 years | 0
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Plasma Membrane Epidermal Growth Factor Receptor (EGFR) Expression, Measured by VECTRA Imaging
Description: An increase of at least 25% from baseline to post-dasatinib treatment will be considered significant. VECTRA is an automated pathology imaging system used to detect biomarkers in samples.
Time Frame: 7-10 days
Measure: Mean (Full Range); unit: percentage plasma EGFR
Arm/Group | Dasatinib 100mg
Number analyzed (Participants) | 5
percentage plasma EGFR
  Baseline | 0.54 [0.43 to 0.61]
  After Treatment | 0.40 [0.00 to 0.77]

2. Secondary Outcome: Number of Treatment-emergent Adverse Events [Safety and Tolerability] up to 4 Weeks
Description: Safety and tolerability of dasatinib in participants with operable Triple negative breast cancer (TNBC) will be based on NCI Adverse Events (AE) Version 4.0 and will be assessed by frequency tables. AEs were collected on day 1 of treatment and a minimum of 14 days after the last dose. AEs reported here were ranked as either possibly related, probably related, or definitely related to the study intervention. All AEs (including not related and unlikely related) are summarized in the AE section.
Time Frame: Up to 4 weeks
Measure: Number; unit: adverse events
Units Other Than Participants: adverse events
Arm/Group | Dasatinib 100mg
Number analyzed (Participants) | 5
Number analyzed (adverse events) | 14
adverse events
  Fatigue | 4
  Anemia | 2
  Creatinine Increase | 1
  Low E-GFR | 1
  Nausea | 1
  Insomnia | 1
  Body Aches | 1
  Constipation | 1
  Headache | 1
  Dyspepsia | 1

3. Secondary Outcome: Number of Participants With Pathologic Complete Response (pCR)
Description: Examine pCR rates to standard neoadjuvant chemotherapy in nuclear Epidermal Growth Factor Receptor (nEGFR) + TNBC. pCR will be defined as ypT0 ypNO (absence of cancer in breast tissue and lymph nodes) an assessed by the investigator.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib 100mg
Number analyzed (Participants) | 5
Participants | 1

4. Secondary Outcome: Number of Participants With No Evidence of Disease (NED) at Long-term Follow up
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib 100mg
Number analyzed (Participants) | 5
Participants
  NED at 16 months (subsequently lost to follow up) | 1
  NED at 24 months | 4

ADVERSE EVENTS:
Time Frame: up to 4 weeks - see limitations and caveats
Arm/Group | Dasatinib 100mg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100mg (N=5)
Neutrophil Count Decreased (Investigations) | 1 (1) — Characterized as unlikely related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100mg (N=5)
Fatigue (General disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine Increase (Investigations) | 1 (1)
Low eGFR (Investigations) | 1 (1) — estimated glomerular filtration rate (eGFR)
Insomnia (Psychiatric disorders) | 1 (1)
Body Aches (General disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
White Blood Cell Count Decreased (Investigations) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
AST increased (Investigations) | 1 (1) — Aspartate aminotransferase (AST)
Proteinuria (Renal and urinary disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Statistical analyses were not completed for this study as it was not powered for meaningful results. Study was terminated early due to pandemic related enrollment issues, participants moved on to other therapies compromising intervention-relevant long term AE follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02720185/Prot_SAP_000.pdf